CLINICAL TRIAL: NCT06141070
Title: Addition of Hypofractionated High Dose Radiation in Oligometastatic Disease - An Open Label Randomized Phase III Trial Comparing Up-front Radiation in Oligometastatic Non-small Cell Lung Cancer (NSCLC) and Systemic Treatment With Systemic Treatment Alone
Brief Title: Addition of Hypofractionated High Dose Radiation in Oligometastatic Disease
Acronym: ANDROMEDA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The ANDROMEDA trial
Record Dates: First submitted 2023-11-13; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A, standard systemic therapy (Active Comparator): Standard systemic chemoimmunotherapy
  Interventions: Drug: Standard systemic therapy
- B, Radiotherapy + systemic therapy (Experimental): Standard systemic chemoimmunotherapy and radiation to all known lesions
  Interventions: Other: Standard systemic therapy + radiotherapy

INTERVENTIONS:
Other: Standard systemic therapy + radiotherapy — Combined systemic therapy + radiation
  Arms: B, Radiotherapy + systemic therapy
Drug: Standard systemic therapy — Chemoimmunotherapy or immunotherapy
  Arms: A, standard systemic therapy

SUMMARY:
This is a 2:1 randomized multicentre open label phase III study of radiation combined with standard systemic treatment compared with systemic treatment alone in oligometastatic (≤5 metastases) NSCLC. Stratification factors: performance status, gender and systemic strategy. The systemic treatment consists of chemotherapy/chemoimmunotherapy or immunotherapy and is given according to local practice. During the first 3 months of systemic treatment, aiming to start around the 2nd cycle is radiotherapy delivered to all known lesions. Preferably with SBRT /SRT/SRS but conventional radiotherapy may also be used. After the first three cycles of systemic treatment, the patients are assessed, and after four cycles, they are continuing maintenance therapy if indicated. The patients are followed with radiology every three months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject prior to performing any protocol- related procedures, including screening procedures

  * Histological or cytological diagnosis of NSCLC
  * Stage IV disease with ≤5 metastases (not including primary tumour or mediastinal nodes, N1-N3)
  * Patient deemed fit for first line chemoimmunotherapy, immunotherapy or chemotherapy
  * Extra-thoracic metastases accessible for stereotactic body radiotherapy (SBRT)
  * Thoracic tumour(s) accessible for SBRT or conventional radiotherapy
  * Received no prior systemic treatment or radiation therapy for NSCLC (previous adjuvant systemic therapy is allowed)
  * Age > 18 years at time of study entry, no upper age limit
  * WHO performance status 0-2
  * Adequate normal organ and marrow function Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal subjects.

    * Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* • Solitary brain lesion or contralateral lung lesion as the only distant metastasis

  * Participation in another clinical study with an investigational product during the last 4 weeks
  * Patients with EGFR+, ALK+, ROS1+ disease or any other genetic alteration that would result in a TKI based first line treatment (i.e. first line treatment not being chemoimmuno- or immunotherapy)
  * Malignant pleural fluid, or ascites (malignant cells or clinical judgement) or excessive fluid hampering radiation according to protocol
  * Leptomeningeal disease
  * Pulmonary fibrosis making protocol stipulated treatment hazardous (low grade radiologic findings are allowed as assessed by the investigator)
  * Not deemed fit for standard first line systemic therapy
  * Second primary residual malignancy. Other malignancy diagnosed and treated > 2 years ago without relapse and deemed to have a low likelihood of relapse is allowed. (Carcinoma in situ of the cervix or adequately treated basal cell carcinoma of the skin < 2 years are allowed, as is other low-grade malignancy with low likelihood of becoming metastatic or impact on survival e.g. low-grade prostate cancer not in need of treatment)
  * Female subjects who are pregnant or breastfeeding or male or female subjects of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of systemic therapy
  * Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of death from any cause, whichever came first, assessed up to 60 months
  Time to death

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization until the date of first documented systemic progression or date of death from any cause, whichever came first, assessed up to 60 months
  Time to progressive disease or death
Local control (LC) | At 12 months after randomization
  Percentage complete, partial remission or stable disease

CONTACTS AND LOCATIONS:
Locations (6):
- Sweden (6):
  - Dept of Oncology, Gothenburg
  - Dept of pulmonary medicine, Linköping
  - Dept of pulmonary medicine, Lund
  - Dept of Oncology, Stockholm
  - Dept. of Oncology, Umeå
  - Dept. of Oncology, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided